CLINICAL TRIAL: NCT07121894
Title: Ketogenic Intervention for Bipolar Depression: An Open-Label Trial Guiding Clinical Implementation (KETO-MAYO)
Brief Title: Ketogenic Intervention for Bipolar Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kyla M. Lara-Breitinger, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-013228
Record Dates: First submitted 2025-07-18; First posted 2025-08-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet (Experimental): Patients diagnosed with bipolar disorder and experiencing depression or depressive symptoms.
  Interventions: Behavioral: Ketogenic Diet

INTERVENTIONS:
Behavioral: Ketogenic Diet — Participants will initiate a modified ketogenic diet under structured, intensive guidance. Simultaneously, participants will attend weekly behavioral support interviews with a psychiatrist to monitor mental health and mood stability.

SUMMARY:
The purpose of this study is to assess the clinical correlates of therapeutic precision ketosis in bipolar depression and to evaluate the cardiometabolic correlates associated with therapeutic precision ketosis in bipolar depression.

ELIGIBILITY:
Inclusion Criteria

* Age 18-50 years
* Willingness to change the current diet to a high fat, low carbohydrate diet
* Diagnosis of bipolar I or II disorder, or BP schizoaffective Disorder by DSM-IV (SCID- confirmed). If a participant has already completed a structured diagnostic interview within the last 2 years or in any of the Department of Psychiatry and Psychology Mood Unit studies, existing SCID results can be used for this study; thus, they will not be required to repeat the SCID assessment. If a structured diagnostic interview was completed more than 2 years ago, the current mood state sections of the SCID must be repeated to ensure accuracy of current mood state assessment.
* Depressive symptom severity of at least mild (MADRS > 6) with steady and stable (ie, at least 2 weeks) mood stabilization (eg, lithium, valproate, lamotrigine, carbamazepine/oxcarbamazepine, and/or atypical antipsychotic therapy) and non-psychotropic medication.
* Urine drug screen is negative except for allowable drugs that they have been prescribed, such as benzodiazepines.
* Pregnancy test is negative.
* Established birth control practice for sexually active individuals.
* Medical comorbidity is stable (hypertension, T2D, gout - uric acid in normal limits).

Exclusion Criteria:

* No access to smartphone or internet (unless provided by sponsor)
* Inability to provide written, voluntary, informed consent and pass (80%) comprehension assessment related to study goals, risks, and benefits.
* Structured clinical interview confirmation of schizophrenia or presence of psychotic symptoms (both SCID and YMRS question 8>5).
* Clinical diagnosis of personality disorder that, upon review by the study psychiatrist, of all available information (SCID, electronic health record), is the primary psychiatric diagnosis.
* Mixed symptoms of depression defined as a YMRS ≥12 (i.e., hypomania).
* Active suicidal ideation as defined by MADRS score >4 on question #10 or Columbia Suicide Severity Scale (C-SSRS), yes response to Question #4 (ideation, intent, but no plan) or Question #5 (ideation, intent, and plan).
* Any current drug and alcohol use disorder (excluding nicotine); complete (not partial) remission ≥3 months.
* Positive toxicology screen for cannabis and cannabis use disorder by structured clinical interview. Participants who use cannabis for recreational or medicinal purposes and fail the toxicology screen can potentially be included if the Cannabis Use Disorder Identification Test (CUDIT-R) score is < 12.
* Currently undergoing ECT, transcranial magnetic stimulation, or deep brain stimulation as an acute or maintenance treatment. Maintenance vagal nerve stimulation is allowed if the placement of device is > 1 year.
* Current involuntary psychiatric hospitalization.
* Already in ketosis or on a medication that causes acidosis, such as carbonic anhydrase inhibitors (e.g., acetazolamide "Diamox" and topiramate).
* BMI < 18.5; (m) baseline LDL-c > 190.
* Any active or unstable medical condition judged by the principal investigator as conferring significant medical risk to allow inclusion in the study, such as active severe infection.
* Acute pancreatitis or history of lipid-associated pancreatitis.
* Type I diabetes.
* SGLT2 inhibitor use
* Rare inborn errors of metabolism affecting fatty acid processing (typically diagnosed in infancy or, rarely, adolescence), such as Pyruvate carboxylase deficiency and Porphyria
* Primary carnitine deficiency
* Chronic renal failure, significant renal disease defined as creatinine clearance <30 or in dialysis.
* Severe vitamin D deficiency (serum levels of 25-hydroxyvitamin D [25(OH)D] < 12 ng/mL or 30 nMol/L).
* A diagnosis of osteopenia, defined as a bone mineral density (BMD) T-score between -1.0 and -2.5 on a dual-energy X-ray absorptiometry (DEXA) scan or with a history of fragility fractures
* Clinically significant laboratory test abnormality
* Anticipated elective surgical procedure within the next 18 weeks
* Family history of premature coronary artery disease defined as atherosclerotic cardiovascular events (e.g., heart attack, stroke) before 55 and 65 years of age in male and female first-degree relatives, respectively.
* History of familial hypercholesterolemia (note -current or start of statin or lipid-lowering drug as part of clinical care is not an exclusion provided managed by a primary care provider) or LDL-C>190 mg/dl (or LDL>160 mg/dl if on lipid lowering therapy) or triglycerides>500 mg/dl.
* History of coronary disease or coronary calcifications or coronary stenosis found in invasive cardiac catheterization or imaging.
* History of ischemic stroke or carotid plaque found on baseline common carotid intima-media thickness (IMT) ultrasound.
* History of peripheral atherosclerotic arterial disease or any other form of clinical atherosclerosis.
* History or current diagnosis of respiratory failure defined as a PaO₂ < 60 mmHg or SpO₂ < 90% on room air or any condition leading to clinically significant respiratory impairment
* History or current diagnosis of liver failure or chronic liver disease with significant impairment, defined as ALT or AST > 5 times the upper limit of normal, or total bilirubin > 3 mg/dL.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | Baseline, 6 months
  Measured using the Quick Inventory for Depressive Symptomatology Clinician Rated (QIDS-C), a 16-item clinician rating, each rated on a four-point Likert scale (0-3). The total score ranges from 0 to 27. The QIDS-C is scored by summing the responses to the 16 items, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Response and Remission Rates | Baseline, 6 months
  Measured using the Montgomery-Asberg Depression Rating Scale (MADRS), with response defined as a ≥50% reduction from baseline symptoms and remission as a score <10, providing complementary measures of symptom improvement. MADRS is a 10-item observer rating scale assessing symptoms of depression. The MADRS will be used to assess depression severity, exclude patients with suicidal ideation scoring > 4 on question #10 and measure % of patients achieving remission defined as a MADRS < 10.
Percentage of clinically significant improvement | Baseline, 6 months
  The proportion of participants rated as "much improved" or "very much improved" on the Clinical Global Impression for Bipolar Disorder (CGI-BP) scale. CGI-BP is a specialized tool for assessing the severity, treatment response, and efficacy of interventions in bipolar disorder. It addresses the unique features of the disorder by evaluating manic and depressive episodes separately. It consists of three components: Severity of Illness (CGI-BP-S), Global Improvement (CGI-BP-I), which tracks changes from baseline; and Efficacy Index (CGI-BP-E), which assesses treatment benefits relative to side effects.
Change in anxiety symptoms | Baseline, 6 months
  Measured using the General Anxiety Disorder 7 (GAD-7), a 7-item self-report questionnaire used to measure the severity of generalized anxiety symptoms over the past two weeks. Each item is scored on a 4-point Likert scale (0 = "Not at all" to 3 = "Nearly every day"), with a total score ranging from 0 to 21. Higher scores indicate greater anxiety severity
Prevalence rate of disordered eating | 6 months
  Measured using the Eating Disorder Diagnostic Scale (EDDS), a standardized measure designed to assess symptoms of eating disorders. It quantifies symptom severity and provides a diagnostic algorithm based on threshold scores that indicate probable diagnoses and subthreshold levels of disordered eating. The EDDS includes 22 items that evaluate key behaviors and cognitive symptoms associated with eating disorders.
Change in psychosocial functioning | Baseline, 6 months
  Measured using the Functioning Assessment Short Test (FAST),a short, simple interview-administered instrument for patients with psychiatric disorders to assess functional recovery. The psychometric properties of this test enable it to detect differences between euthymic and acute patients with bipolar disorder. The total FAST score is the sum of each item. Lower scores indicate good functioning, while higher scores indicate increased impairment.
Change in well-being | Baseline, 6 months
  Measured using the Well-Being Index (WHO-5), a self-report instrument measuring mental well-being. It consists of five statements relating to the past two weeks. Each statement is rated on a 6-point scale, with higher scores indicating better mental well-being.
Change in insulin resistance | Baseline, 6 months
  Insulin resistance will be assessed using calculated Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) from fasting glucose and insulin levels.
Change in mitochondrial function | Baseline, 6 months
  Assessed by evaluating baseline-to-endpoint changes in mitochondrial metabolites, measured using the MMPP test developed at Mayo Clinic.
Change in serum levels of high sensitivity C-reactive protein (CRP) | Baseline, 6 months
  High sensitivity C-reactive protein (CRP) is an acute-phase protein produced by the liver in response to systemic inflammation and is widely used as a biomarker of inflammation. These changes will be analyzed in conjunction with daily ketone body measurements, providing an index of ketosis.
Change in subclinical vascular health | Baseline, 6 months
  Assessed by changes in key vascular function and structure indicators. This includes detailed assessments of lipid profiles, focusing on biomarkers such as apolipoprotein B and advanced high-resolution lipoprotein subfraction profiling.
Change in interleukin-6 IL-6 | Baseline, 6 months
  Interleukin-6 (IL-6) is a cytokine involved in immune response and inflammation. These changes will be analyzed in conjunction with daily ketone body measurements, providing an index of ketosis, and mood state assessments to explore potential correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Kyla M. Lara-Breitinger, MD, Principal Investigator — Mayo Clinic; Mark Frye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials